CLINICAL TRIAL: NCT04375865
Title: A Phase I Clinical Trial to Evaluate the Pharmacokinetic Interactions and Safety Between AD-2111 and AD-2112 in Healthy Adult Subjects
Brief Title: Evaluating the Pharmacokinetic Interactions and Safety Between AD-2111 and AD-2112
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Addpharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: AD-211DDI
Record Dates: First submitted 2020-04-27; First posted 2020-05-06 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Treatment A (Experimental): Period1: Celecoxib 200mg Period2: Tramadol 150mg Period3: Celecoxib 200mg + Tramadol 150mg
  Interventions: Drug: AD-2111; Drug: AD-2112
- Treatment B (Experimental): Period1: Celecoxib 200mg Period2: Celecoxib 200mg + Tramadol 150mg Period3: Tramadol 150mg
  Interventions: Drug: AD-2111; Drug: AD-2112
- Treatment C (Experimental): Period1: Tramadol 150mg Period2: Celecoxib 200mg Period3: Celecoxib 200mg + Tramadol 150mg
  Interventions: Drug: AD-2111; Drug: AD-2112
- Treatment D (Experimental): Period1: Tramadol 150mg Period2: Celecoxib 200mg + Tramadol 150mg Period3: Celecoxib 200mg
  Interventions: Drug: AD-2111; Drug: AD-2112
- Treatment E (Experimental): Period1: Celecoxib 200mg + Tramadol 150mg Period2: Celecoxib 200mg Period3: Tramadol 150mg
  Interventions: Drug: AD-2111; Drug: AD-2112
- Treatment F (Active Comparator): Period1: Celecoxib 200mg + Tramadol 150mg Period2: Tramadol 150mg Period3: Celecoxib 200mg
  Interventions: Drug: AD-2111; Drug: AD-2112

INTERVENTIONS:
Drug: AD-2111 — celecoxib 200mg
Drug: AD-2112 — Tramadol 150mg

SUMMARY:
A phase I clinical trial to evaluate the pharmacokinetic interactions and safety between AD-2111 and AD-2112

DETAILED DESCRIPTION:
Purpose: pharmacokinetic interactions and safety of AD-2111 and AD-2112 in healthy adult volunteers Condition or disease : Pain Intervention/treatment Drug : AD-2111(Celecoxib 200mg), AD-2112(Tramadol 150mg) Phase : Phase 1

ELIGIBILITY:
Inclusion Criteria:

* Healthy Adult aged 19 and more at the time of screening visit
* Body mass index (BMI) between 18.5 kg/m2 and 27.0 kg/m2 at the time of screening visit

Exclusion Criteria:

* As a result of laboratory tests, the following figures: ALT or AST or total bilirubin > 1.5 times upper limit of normal range
* As a result of laboratory tests, the following figures: Creatinine clearance < 80mL/min

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-05-30 (Actual); Primary Completion 2020-07-16 (Actual); Study Completion 2020-07-16 (Actual)

PRIMARY OUTCOMES:
Area under the curve in time plot (AUCt) | pre-dose to 72 hours
  AUCt of the total ingredient of Celecoxib, Tramadol
Peak Plasma Concentration (Cmax) | pre-dose to 72 hours
  Cmax of the total ingredient of Celecoxib, Tramadol

SECONDARY OUTCOMES:
Area under the curve in time plot (AUCinf) | pre-dose to 72 hours
  AUCinf of the total ingredient of Celecoxib, Tramadol, O-desmethyltramadol
Time to reach Cmax(Tmax) | pre-dose to 72 hours
  Tmax of the total ingredient of Celecoxib, Tramadol, O-desmethyltramadol
Effective half-life(t1/2) | pre-dose to 72 hours
  t1/2 of the total ingredient of Celecoxib, Tramadol, O-desmethyltramadol
Clearance(CL/F) | pre-dose to 72 hours
  CL/F of the total ingredient of Celecoxib, Tramadol, O-desmethyltramadol
Volume of distribution(Vd/F) | pre-dose to 72 hours
  Vd/F of the total ingredient of Celecoxib, Tramadol, O-desmethyltramadol
Area under the curve in time plot (AUCt) of O-desmethyltramadol | pre-dose to 72 hours
  AUCt of the total ingredient of O-desmethyltramadol
Peak Plasma Concentration (Cmax) of O-desmethyltramadol | pre-dose to 72 hours
  Cmax of the total ingredient of O-desmethyltramadol

CONTACTS AND LOCATIONS:
Overall Officials: Young-Ran Yoon, M.D., Ph.D, Principal Investigator — Kyungpook National University Hospital
Locations (1):
- Kyungpook National University Hospital, Daegu, South Korea